CLINICAL TRIAL: NCT03717623
Title: Pharmacokinetics Study of Posaconazole in Haematology Patients Receiving Standard of Care Treatment With Oral Posaconazole Prophylaxis for Invasive Fungal Infection
Brief Title: Posaconazole Pharmacokinetics in Patients Receiving Chemotherapy or Stem Cell Transplants
Acronym: POPULAR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017.105
Record Dates: First submitted 2018-10-10; First posted 2018-10-24 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Posaconazole; Pharmacokinetics; Invasive Candidiases; Invasive Aspergillosis; Invasive Mycosis; Fungal Infection; Prophylaxis
MeSH Terms: conditions — Candidiasis, Invasive; Invasive Fungal Infections; Mycoses | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Posaconazole prophylaxis (Experimental): Blood samples will be taken from participants undergoing cancer treatment and receiving Posaconazole prophylaxis. The samples will be used for Posaconazole pharmacokinetics study.
  Interventions: Drug: Posaconazole pharmacokinetics

INTERVENTIONS:
Drug: Posaconazole pharmacokinetics — Blood samples will be collected on Days 7, 14 and 21 from the onset of Posaconazole prophylactic treatment If significant diarrhoea occurs, additional blood samples will be collected twice weekly until symptoms resolve. All blood samples will be used for Posaconazole pharmacokinetics study.
  Other Names: Blood sampling

SUMMARY:
The purpose of the study is to investigate the pharmacokinetics of oral dosage of Posaconazole which is routinely administered as a standard care prophylaxis for patients undergoing cancer treatments.

DETAILED DESCRIPTION:
Participants receiving Posaconazole prophylaxis for invasive fungal infection while undergoing cancer treatment will be required to sign an informed consent and donate blood samples for the study. Posaconazole is routinely administered as a prophylaxis using the oral tablet formulation (300mg once daily) as a standard care. Each prophylaxis course-duration will be defined according to local policy at each hospital. In general, Posaconazole prophylaxis commences prior to or with induction or consolidation chemotherapy in AML/MDS patients and continues until neutrophil recovery. In allo-HSCT setting, Posaconazole prophylaxis routinely commences on the day of transplant or with conditioning chemotherapy and continues for approximately 3 months after transplant, except in patients with initiation of intensive immunosuppression after diagnosis of acute or chronic GVHD, administration will go for at least 16 weeks or until prednisolone dose is less than 10mg per day, whichever is later. If patients are suspected or have proven malabsorption or are required to switch to an alternative antifungal agent such as in the case of suspected invasive fungal infection or Posaconazole toxicity, a switch to intravenous formulation of Posaconazole will take place.

Blood samples will be collected on Days 7, 14 and 21 from the onset of Posaconazole prophylactic treatment. If significant diarrhoea occurs, additional blood samples will be collected twice weekly until symptoms resolve, with the first sample being taken 3 days after the onset of diarrhoea. If gastrointestinal absorption is considered inadequate or invasive fungal infection is suspected and patients are switched either to IV antifungal prophylaxis or antifungal treatment as part of their standard care, a blood sample will be collected 20-24 hours after the last oral Posaconazole dose. Study participants will be followed up with respect to clinical data collection during the blood sample collection period and for up to 7 days after the last dose of Posaconazole for invasive fungal infection follow-up, and for the entire antifungal prescribing period (prophylaxis and/or treatment). Participants with diagnosed invasive fungal infection will be followed up to 30-days post-diagnosis with respect to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old) haematology patients receiving Posaconazole prophylaxis in the inpatient setting as standard of care.
* Able to give informed consent.

Exclusion Criteria:

* Unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pre-dose plasma Posaconazole concentrations | On days 7, 14 and 21 of Posaconazole prophylaxis course, when significant diarrhea occurs, when active gastrointestinal graft versus host disease occurs.
  The median interquartile range pre-dose plasma Posaconazole concentrations equal or greater than 0.7 mg/L will be assessed.

SECONDARY OUTCOMES:
Clinical symptoms affecting plasma Posaconazole concentrations. | At Screening, Days 7, 14 and 21, and 72 hours after onset of diarrhoea, and when invasive fungal infection occurs.
  Observed association between concurrent patient factors with change in plasma Posaconazole concentrations.
The number/proportion of patients achieving desirable pre-dose plasma Posaconazole concentrations. | On days 7, 14 and 21 of Posaconazole prophylaxis course, when significant diarrhea occurs, when active gastrointestinal graft versus host disease occurs.
  The number/proportion of patients achieving pre-dose plasma Posaconazole concentrations greater or equal to 0.7 mg/L will be assessed.
Effects of diarrhea on plasma Posaconazole concentration | When diarrhea occurs during Posaconazole prophylaxis on Days 1 to 21.
  Correlation between the presence/extent of diarrhea with change in plasma Posaconazole concentrations.
Alteration in prophylaxis due to Posaconazole-attributed toxicities. | When change in or cessation of oral Posaconazole prophylaxis occurs during Day 1 to Day 21.
  Frequency of Posaconazole-attributed toxicities resulting in dose changes or cessation of prophylaxis will be noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Melbourne Health, Parkville, Victoria, Australia